CLINICAL TRIAL: NCT01731054
Title: Noninvasive Assessment Of Renal Activity And Damage Using Renal Functional MRI In Normal Healthy Volunteers And Subjects With Lupus Nephritis
Brief Title: Functional MRI in Lupus Nephritis
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 999LE002
Record Dates: First submitted 2012-11-08; First posted 2012-11-21 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-03

CONDITIONS: Healthy; Lupus Nephritis
Keywords: lupus nephritis; normal healthy volunteer; MRI
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Samples, Urine samples and Renal biopsy tissue samples.
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objectives of the study are as follows: To develop and optimize a renal functional magnetic resonance imaging (MRI) protocol consisting of Diffusion-Weighted Magnetic Resonance Imaging (DW-MRI), Blood-Oxygen- Level-Dependent MRI (BOLD-MRI), Arterial Spin Labeling MRI (ASL-MRI), Phase Contrast MRI (PC-MRI), and T1rho-MRI; To compare renal functional MRI cross-sectional readouts between normal healthy volunteers (NHV) and lupus nephritis (LN) participants.

The secondary objectives of this study are as follows: Explore whether renal functional MRI techniques discriminate between renal inflammatory activity and damage in lupus nephritis (LN); To examine whether renal functional MRI measurements correlate with laboratory features of renal involvement and renal function in participants with lupus nephritis (LN).

ELIGIBILITY:
Key Inclusion Criteria:

* Must have a documented diagnosis of systemic lupus erythematosus (SLE) according to current American Academy of Rheumatology (ACR) criteria. At least 4 American Academy of Rheumatology (ACR) criteria must be documented, 1 of which must be a positive antinuclear antibody (ANA), anti-Sm, or anti-double stranded DNA antibody.
* Must have a standard of care renal biopsy for lupus nephritis performed or scheduled within +/-7 days of Day 1.

Key Exclusion Criteria:

* Has a metal device affected by magnetic resonance imaging (MRI )(e.g., any type of electronic, mechanical, or magnetic implant; cardiac pacemaker; aneurysm clips; implanted cardiac defibrillator), or has potential ferromagnetic foreign body (metal slivers, metal shavings, other metal objects) that would be a contraindication for magnetic resonance imaging (MRI).
* History of renal transplant.
* Subjects with uncontrolled diabetes or other condition that may result in significant renal disease.

NOTE: Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Primary care clinic, community sample. 30 Normal Healthy Volunteers 30 Participants with documented diagnosis of Lupus Nephritis
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The test-retest reliability and sensitivity of renal functional magnetic resonance imaging (MRI) measurements to detect renal inflammatory activity or damage in normal healthy volunteers (NHV) and participants with lupus nephritis (LN). | Day 1
The mean difference between normal healthy volunteers (NHV) and lupus nephiritis (LN) groups in renal structural and functional magnetic resonance imaging (MRI) measurements. | Within7 days of renal biopsy

SECONDARY OUTCOMES:
Correlation between histological renal activity and chronicity scores and renal functional magnetic resonance imaging (MRI) measurements in participants with lupus nephritis (LN). | Day 1
Correlation between renal cortical volume and renal functional magnetic resonance imaging (MRI) measurements. | Day 1
Correlation between renal functional magnetic resonance imaging (MRI) measurements and renal function as assessed by estimated glomerular filtration rate (eGFR) using Modification of Diet in Renal Disease (MDRD) formula. | Day 1
Correlation between renal functional magnetic resonance imaging (MRI) measurements and proteinuria. | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (4):
- United States (4):
  - Research Site, Los Angelos, California
  - Research Site, Torrance, California
  - Research Site, The Bronx, New York
  - Research Site, Columbus, Ohio